CLINICAL TRIAL: NCT00758407
Title: Placebo Controlled Double Blind Study With Methylphenidate in Treatment of Adults With Cancer-Related Fatigue
Brief Title: Methylphenidate Treatment of Cancer-Related Fatigue
Acronym: EMF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Responsible Party: Dr. Armin Engels, Medical Advisor, Medice Arzneimittel Pütter GmbH & Co KG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6520-9959-02
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Cancer-related Fatigue
Keywords: Fatigue, Cancer, Methylphenidate,
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Methylphenidate hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate hydrochloride — sustained release, dosage according to an individual titration schedule
  Arms: 1
Drug: Placebo — dosage according to an individual titration schedule
  Arms: 2

SUMMARY:
The purpose of this randomized controlled clinical trial is to investigate the efficacy and safety of methylphenidate in patients with fatigue caused by cancer.

ELIGIBILITY:
Inclusion Criteria:

* history of Cancer
* MFI >40
* Karnofsky Index >=70
* outpatient
* patient are able to give informed consent

Exclusion Criteria:

* treatment with psychostimulants in the past two weeks before screening
* active tumor disease
* depression (HADS >10)
* cachexia (BMI <18kg/m2)
* clinically relevant kidney disorders
* clinically relevant liver disorder
* pathological ECG-finding
* high blood pressure
* occlusive arterial disease
* angina pectoris
* cardiac arrhythmias
* CHD
* post heart-attack status
* post stroke status
* known elevated intra-ocular pressure
* known enlarged prostates
* latent and manifest hyperthyreosis
* alcohol, medication or drug dependency in the past six months or manifest drug abuse
* participation in a clinical study within the past 30 days
* participation in this study at an earlier point in time
* simultaneous participation in another clinical trial
* women of child-bearing age without adequate contraception (contraceptives, intrauterine device , no sexual intercourse)
* pregnancy (positive pregnancy test) or lactation period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2006-08; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
General Fatigue measured by the Multidimensional Fatigue Inventory (Subscale General Fatigue) | 6 weeks

SECONDARY OUTCOMES:
Quality of Life (EORTC-QLQ C30) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Heim, Prof., Principal Investigator — Sonnenbergklinik, Hardstr. 13, D-37242 Bad Sooden-Allendorf
Locations (6):
- Germany (6):
  - Sonnenbergklinik, Bad Sooden-Allendorf
  - Dr. J.-U. Rüffer, Cologne
  - Praxis Dr. Lathan, Dortmund
  - Praxis Dr. Verpoort - Dr. Zeller, Hamburg
  - Medizinische Fakultät der Universität Leipzig, Leipzig
  - Medizinisches Versorgungszentrum - MOP, München